CLINICAL TRIAL: NCT00307918
Title: Acupuncture Treatment for Elevated Intraocular Pressure: A Pilot Study
Brief Title: Acupuncture for Elevated Intraocular Pressure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of patients
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP GL 01 06 CTIL
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-09

CONDITIONS: Elevated Intraocular Pressure
Keywords: acupuncture, intraocular pressure, glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — Acupuncture Therapy

INTERVENTIONS:
Device: acupuncture

SUMMARY:
Glaucoma is the leading cause of irreversible blindness in the world, resulting from progressive axonal destruction of the optic nerve. Primary open-angle glaucoma is the most common form, and it is usually painless with insidious onset. Conventional treatment is focused on lowering intraocular pressure (IOP), the one risk factor that can be modified, which has been demonstrated to protect against further damage to the optic-nerve head. Acupuncture is an ancient treatment which has been found to be beneficial for many ailments, and may reduce IOP. We propose a pilot study to evaluate whether acupuncture is an effective and safe modality for reducing elevated IOP in patients with open angle glaucoma and primary ocular hypertension. Patients with elevated IOP on tonometric measurement (20mmHg < IOP < 30mmHg) will be treated twice-weekly with a standardized (as opposed to individualized) acupuncture treatment. Treatment will last for four-weeks (for a total of 8 treatments), and patients will be evaluated for IOP diurnal curves at 2 weeks (4 treatment), 4 weeks (end of treatment ) and then 4 weeks following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

patients of either gender; age 21 years and older; intraocular pressure equal/greater than 20mmHg, equal/less than 30mmHg; ability to comply with study protocol

Exclusion Criteria:

patients with secondary or closed-angle glaucoma; patients with a history of laser or other surgical treatment of glaucoma; patients displaying symptoms of depression, anxiety or psychosis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Intraocular pressure curves.

SECONDARY OUTCOMES:
safety of acupuncture treatment

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Dept. of Ophthalmology, Shaare Zedek Medical Center, Jerusalem, Israel